CLINICAL TRIAL: NCT00868127
Title: An Open-Label Extension Study to Evaluate the Safety and Tolerability of Lapaquistat Acetate in Subjects With Hypercholesterolemia
Brief Title: Safety of Lapaquistat Acetate in Subjects With Hypercholesterolemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 01-04-TL-475-010; U1111-1122-8368 (Registry Identifier: WHO)
Record Dates: First submitted 2009-03-18; First posted 2009-03-24 (Estimated); Last update posted 2012-05-24 (Estimated); Status verified 2012-05

CONDITIONS: Hypercholesterolemia
Keywords: Hyperlipidemia; Drug Therapy; Dyslipidemia
MeSH Terms: conditions — Hypercholesterolemia; Hyperlipidemias; Dyslipidemias | interventions — 1-((1-(3-acetoxy-2,2-dimethylpropyl)-7-chloro-5-(2,3-dimethoxyphenyl)-2-oxo-1,2,3,5-tetrahydro-4,1-benzoxazepin-3-yl)acetyl)piperidine-4-acetic acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Lapaquistat Acetate 100 mg QD (Experimental)
  Interventions: Drug: Lapaquistat acetate
- Lapaquistat Acetate 100 mg QD + Added Therapy (Experimental)
  Interventions: Drug: Lapaquistat acetate and additional lipid-lowering therapy

INTERVENTIONS:
Drug: Lapaquistat acetate — Participants from 01-04-TL-475-008 Monotherapy Study:
  Lapaquistat acetate 100 mg, tablets, orally, once daily for up to 48 weeks.
  Other Names: TAK-475
  Arms: Lapaquistat Acetate 100 mg QD
Drug: Lapaquistat acetate and additional lipid-lowering therapy — Participants from 01-04-TL-475-009 Atorvastatin Add-on Study:
  Lapaquistat acetate 100 mg, tablets, orally, once daily and current Atorvastatin therapy for up to 4 weeks.
  Then, Lapaquistat 100 mg, tablets, orally, once daily and dose adjustment of Atorvastatin OR additional companion lipid-lowering therapy as needed for target LDL-C for up to 42 weeks.
  Other Names: TAK-475
  Arms: Lapaquistat Acetate 100 mg QD + Added Therapy

SUMMARY:
The purpose of this study is to determine the long-term safety of lapaquistat acetate, once daily (QD), as monotherapy or in combination with other lipid-lowering agents in Subjects with Hypercholesterolemia.

DETAILED DESCRIPTION:
Elevated plasma cholesterol (hypercholesterolemia) and various other plasma lipid imbalances (dyslipidemias) are major risk factors for coronary heart disease. Normally, the balance among cholesterol synthesis, dietary intake, and degradation is adequate to maintain healthy cholesterol plasma levels. However, in patients with hypercholesterolemia, elevation in low-density lipoprotein cholesterol leads to atherosclerotic deposition of cholesterol in the arterial walls. Consequently, it has been established that lowering the low-density lipoprotein cholesterol plasma concentration effectively reduces cardiovascular morbidity and mortality. As a result of this finding, the National Cholesterol Education Program Adult Treatment Panel III identifies control of low-density lipoprotein cholesterol as essential in the prevention and management of coronary heart disease. Additional lipid risk factors designated by Adult Treatment Panel III include elevated triglycerides, elevated non-high density lipoprotein cholesterol, and low levels of high-density lipoprotein cholesterol. Lipoproteins rich in triglycerides, such as very low-density lipoprotein cholesterol, appear to contribute to atherosclerosis, whereas the apparent protective effect of high-density lipoprotein cholesterol may be limited at low density lipoprotein concentrations.

Lapaquistat acetate is a squalene synthase inhibitor currently under development at Takeda for the treatment of dyslipidemia.

Participants in this study have primary hypercholesterolemia and have completed either the 12-week monotherapy protocol 01-04-TL-475-008 (NCT00143663) or the 24-week atorvastatin add-on study 01-04-TL-475-009 (NCT00143676).

ELIGIBILITY:
Inclusion Criteria:

* Has completed the 01-04-TL-475-008 or 01-04-TL-475-009 study.
* Females of childbearing potential who are sexually active must agree to use a medically accepted means of contraception, and can neither be pregnant nor lactating from Screening throughout the duration of the study.
* Has clinical laboratory evaluations within reference range for the testing laboratory at the previous visit in study 01-04-TL-475-008 or 01-04-TL-475-009 unless the results were deemed not clinically significant by the investigator or sponsor.
* Is willing and able to comply with a standardized low cholesterol diet.
* Is willing to continue taking the protocol-specified companion lipid-altering medication from the previous study (if applicable) for at least the first 4 weeks.

Exclusion Criteria:

* Has an alanine aminotransferase or aspartate aminotransferase level greater than or equal to 3 times the upper limit of normal at the previous visit in the prior study, active liver disease, or jaundice.
* Has serum creatinine greater than or equal to 133 μmol/l at the previous visit in the prior study.
* Has a creatine kinase greater than or equal to 10 times the upper limit of normal at the previous visit in the prior study.
* Has a previous history of cancer that had been in remission for less than 5 years prior to the first dose of study medication. This criterion did not include those subjects with basal cell or Stage 1 squamous cell carcinoma of the skin.
* Has an endocrine disorder, such as Cushing's syndrome, hyperthyroidism, or inappropriately treated hypothyroidism, affecting lipid metabolism.
* Has a positive hepatitis B surface antigen, or hepatitis C virus antibody, as determined by medical history and/or participant's verbal report.
* Has a positive human immunodeficiency virus status or was taking antiretroviral medications, as determined by medical history and/or subject's verbal report.
* Has a known hypersensitivity to lapaquistat acetate.
* Has a history or presence of clinically significant food allergy that prevented them from maintaining Therapeutic Lifestyle Change (or equivalent) diet.
* Has a known homozygous familial hypercholesterolemia or known Type III hyperlipoproteinemia.
* Has fibromyalgia, myopathy, rhabdomyolysis, or unexplained muscle pain.
* Has uncontrolled hypertension at Visit 1.
* Has inflammatory bowel disease or any other malabsorption syndrome or had gastric bypass or any other surgical procedure for weight loss.
* Has a history of drug abuse or a history of alcohol abuse within the past 2 years.
* Has any other serious disease or condition at Visit 1 that may reduce life expectancy, impair successful management according to the protocol, or make the participant unsuitable to receive study medication.
* Is required to take or intends to continue taking any disallowed medication, any prescription medication, herbal treatment or over-the counter medication that may interfere with evaluation of the study medication, including:

  * Orlistat
  * Sibutramine
  * Isotretinoin
  * Tacrolimus
  * Probucol
  * Systemic corticosteroids and androgens
  * Potent cytochrome P-450 3A4 inhibitors
  * Azole antifungal agents
  * Cyclosporine
  * Erythromycin
  * Clarithromycin
  * Human Immunodeficiency Virus protease inhibitors
  * Amiodarone
  * Verapamil
  * Diltiazem
  * Nefazodone
  * Large quantities of grapefruit juice
  * Warfarin
  * Digoxin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2005-12; Primary Completion 2007-07 (Actual); Study Completion 2007-07 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Weeks 2, 4, 8, 12, 24, 36 and 48
Vital Signs | Weeks 2, 4, 8, 12, 24, 36 and 48
Clinical Laboratory Blood Sample for Lipid Panel | Weeks 2, 4, 8, 12, 24, 36 and 48
Clinical Laboratory Serum Chemistries | Weeks 2, 4, 8, 12, 24, 36 and 48
Clinical Laboratory Hematology | Weeks 2, 4, 8, 12, 24, 36 and 48
Clinical Laboratory Serum Human Chorionic Gonadotropin | Weeks 2, 4, 8, 12, 24, 36 and 48
Clinical Laboratory Urinalysis | Weeks 2, 4, 8, 12, 24, 36 and 48
Physical Examination | Week 48
12-lead Electrocardiogram | Week 48
Best Corrected Visual Acuity | Week 48

SECONDARY OUTCOMES:
Percent change from Baseline in calculated Low Density Lipoprotein Cholesterol | Week 48
Percent change from Baseline in calculated Non-High Density Lipoprotein Cholesterol | Week 48
Percent change from Baseline in calculated Total Cholesterol | Week 48
Percent change from Baseline in calculated Triglycerides | Week 48
Percent change from Baseline in calculated High Density Lipoprotein Cholesterol | Week 48
Percent change from Baseline in Derived ratios Total Cholesterol / High Density Lipoprotein Cholesterol and Low Density Lipoprotein Cholesterol / High Density Lipoprotein Cholesterol | Week 48

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda